CLINICAL TRIAL: NCT07215507
Title: Effect of Timing of Physician Rounds on Hospital Experience for High-Risk Antepartum Patients: A Randomized Controlled TrialTiming of Physician Rounds for Antepartum Patients
Brief Title: Timing of Physician Rounds for Antepartum Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Pro00118226
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Physician Rounds; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Rounding (Active Comparator): The current standard of rounding on the Antepartum service involves a preliminarily bedside encounter with patients between 5-7am by a resident +/- medical student before an attending physician-led Antepartum team discussion from 8-9am. The patient is then rounded on for a second time in the late morning by the entire Antepartum team where patient concerns are heard and care plans for the day are relayed/reiterated/cemented.
  Interventions: Behavioral: Standard Rounding
- Discovery Rounding (Experimental): For certain patients with appropriate clinical risk factors, our service has adopted a policy of "discovery rounding". This method involves solely electronic health record chart review prior to the 8am attending-led Antepartum team discussion where the patient's overnight events are "discovered", clinical courses discussed, and daytime plans proposed. "Discovery rounding" consolidates bedside physician-patient encounters to one mid-morning interaction, forgoing early morning disturbances.
  Interventions: Behavioral: Discovery Rounding

INTERVENTIONS:
Behavioral: Discovery Rounding — For certain patients with appropriate clinical risk factors, our service has adopted a policy of "discovery rounding". This method involves solely electronic health record chart review prior to the 8am attending-led Antepartum team discussion where the patient's overnight events are "discovered", clinical courses discussed, and daytime plans proposed. "Discovery rounding" consolidates bedside physician-patient encounters to one mid-morning interaction, forgoing early morning disturbances.
  Arms: Discovery Rounding
Behavioral: Standard Rounding — The current standard of rounding on the Antepartum service involves a preliminarily bedside encounter with patients between 5-7am by a resident +/- medical student before an attending physician-led Antepartum team discussion from 8-9am. The patient is then rounded on for a second time in the late morning by the entire Antepartum team where patient concerns are heard and care plans for the day are relayed/reiterated/cemented.
  Arms: Standard Rounding

SUMMARY:
This study will include patients admitted to the Antepartum service at Duke University Hospital, many of whom are managing high-risk pregnancies that require extended hospital stays and frequent physician interactions. Currently, two rounding methods are used interchangeably for patients who do not have pregnancy or delivery complications that would preclude participation in delayed daytime rounding. This randomized controlled trial will compare two rounding models: the standard model, in which patients receive two rounds (an early morning bedside encounter and a later team discussion), and the intervention model, which consolidates both rounds into a single, later-morning bedside encounter following the team's review of clinical data. The primary objective is to assess whether consolidating physician rounds into a single, later-morning encounter-referred to as discovery rounding-improves patient satisfaction with communication.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women greater than 20 weeks gestation admitted to the antepartum list at Duke University Hospital

Exclusion Criteria:

* Stillbirth
* ICU admission
* Admission to off-service unit
* Active magnesium sulfate administration
* Active severe hypertension or initiation of anti-hypertensive pathway within past 8 hours
* Category II fetal heart rate tracing
* Other pregnancy/delivery complication precluding delayed rounding
* Unstable/unsuitable condition per overnight team or attending physician
* Previously enrolled/on active board >1 day at morning rounds
* Postpartum readmission
* Antepartum admission within the last 4 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of items rated as "Excellent" on the Communication Assessment Tool (CAT) | One of the following timepoints (whichever comes first for that patient); Hospital day 6 or the immediate postpartum period: postpartum day 0 or 1, depending on the time of delivery
  The CAT measures patients' perceptions of physician communication across 15 specific behaviors, such as listening carefully, showing respect, explaining information clearly, and spending sufficient time with the patient. Each item is rated on a 5-point Likert scale ranging from "Poor" to "Excellent." By focusing on the frequency of "Excellent" ratings, the CAT provides a robust, patient-centered measure of the effectiveness and impact of physician communication during hospitalization.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | At the 6 week postpartum visit
  A 10-item self-report questionnaire, validated for both postpartum and antepartum use, in which each item is scored 0-3 (total 0-30), with higher scores indicating greater depressive symptoms and a common cut-off of ≥13 suggesting possible clinical depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Kelly, MD, Study Director — Duke University Hospital; Rachel Wood, MD, Principal Investigator — Duke University Hospital
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No